CLINICAL TRIAL: NCT01984008
Title: A Prospective, Randomized Controlled Clinical Study of the Efficacy and Safety of Bowklean and Klean-Prep With Dulcolax for the Bowel Preparation Prior Colonoscopy
Brief Title: A Study of the Efficacy and Safety of Bowklean and Klean-Prep With Dulcolax for the Bowel Preparation Prior Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universal Integrated Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UIC-BKL-2013
Record Dates: First submitted 2013-10-24; First posted 2013-11-14 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Bowel Preparation Before Colonoscopy
MeSH Terms: interventions — picosulfate sodium; Magnesium Oxide; Citric Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- picosulfate,MgO, citric acid, bowel preparation, powder (Experimental): colonoscopy picosulfate,MgO, citric acid, bowel preparation, powder
  Interventions: Drug: Picosulfate sodium, magnesium oxide, citric acid
- polyethylene glycol, bisacodyl, (Active Comparator): colonoscopy polyethylene glycol,powder bisacodyl,tablet
  Interventions: Drug: Picosulfate sodium, magnesium oxide, citric acid

INTERVENTIONS:
Drug: Picosulfate sodium, magnesium oxide, citric acid

SUMMARY:
The primary objective of this study is to demonstrate that investigation medication (Bowklean) is not less effective than the active comparator (Klean-Prep with Dulcolax), with regards to the overall quality of bowel preparation in subjects undergoing colonoscopy. An additional objective of this study is to collect subject's response to the acceptability and tolerability about bowel preparation and safety information.

After bowel preparation, independent evaluator who is blinded to subject's treatment will evaluate the overall colon cleansing based on Aronchick and Ottawa scale. A total of 600 eligible subjects scheduled to a colonoscopy will be randomly assigned with equal allocation to 1 of 2 treatment groups: "Bowklean" or "Klean-Prep" with Dulcolax. Each subject's participation is expected to be maximally 4 weeks in study duration (up to 3-week screening period followed by one week post colonoscopy).

DETAILED DESCRIPTION:
The objective of this study was to demonstrate that investigational medication (Bowklean) is not less effective than the active comparator (Klean-Prep with Dulcolax), with regards to the overall quality of bowel preparation in subjects undergoing colonoscopy. It was designed to measure the number of subjects whose colons are cleansed successfully.

The primary efficacy endpoint is the percentage of subjects that achieve excellent or good cleansing (success rate) in the Aronchick Scale.

The secondary efficacy variables include:

1. Proportion of successes (excellent, good, or fair) by individual colon segment (ascending, transverse, descending), which are assessed with the Ottawa scale6.
2. Mean bowel preparation score assessed with Ottawa Scale by adding points for the cleansing of three parts of colon and points for amount of fluid in the bowel.
3. Percentage of subject's responses to the acceptability and tolerability

Safety was assessed at each clinic visit by evaluation of the following variables:

1. Percentage of subjects occurred solicited event (nausea, vomiting, chest pain and dizziness) during the preparation.
2. Percentage of subjects with treatment-emergent adverse events during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 20 and 80 years, inclusive.
* Men or non-pregnant women who are scheduled for an elective colonoscopy.
* Subjects should be willing, able to complete the entire procedure and to comply with study instructions.
* Written informed consent obtained prior to study.

Exclusion Criteria:

* Acute surgical abdominal conditions (e.g. acute obstruction or perforation, etc.)
* Active (acute/exacerbation of/severe/uncontrolled) Inflammatory Bowel Disease (IBD)
* Colon disease (history of colonic cancer, toxic megacolon, toxic colitis, idiopathic pseudo- obstruction, hypomotility syndrome)
* Gastrointestinal disorder (active ulcer, outlet obstruction, gastric retention, gastroparesis, ileus)
* Any prior colorectal surgery in the past 3 months, excluding appendectomy, hemorrhoid surgery or prior endoscopic procedures
* History of upper gastrointestinal surgery (gastric resection, gastric banding, gastric by-pass)
* Severe chronic constipation
* Ascites
* Renal insufficiency ((serum creatinine > 1.5 times the upper limit of normal (ULN))creatinine clearance < 30 mL/min)
* Uncontrolled angina and/or Myocardial Infarction (MI) within last 3 months before randomization, Congestive Heart Failure (CHF), or uncontrolled hypertension
* Participation in an investigational study within 60 days prior to receiving study medication
* Any clinically significant laboratory value at screening, including pre-existing electrolyte abnormality, based on clinical history that the Investigator feels may affect the study evaluation
* Hypersensitivity to any ingredient in the study medication

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2014-03-24 (Actual); Study Completion 2014-06-17 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects that achieve excellent or good cleansing (success rate) in the Aronchick Scale. | six months

SECONDARY OUTCOMES:
Proportion of successes (excellent, good, or fair) by individual colon segment (ascending, transverse, descending), which are assessed with the Ottawa scale. | six months

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided